CLINICAL TRIAL: NCT05543356
Title: A Randomised Controlled Trial to Assess the Immunogenicity, Safety and Reactogenicity of a Second Standard Monovalent (Ancestral) or Bivalent Omicron-specific COVID-19 Vaccine Booster Dose (Pfizer-BioNTech or Moderna) in Healthy Adults in Australia.
Brief Title: COVID-19 Fourth Dose Study in Australia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawal of supply of vaccine from one manufacturer
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other); The Peter Doherty Institute for Infection and Immunity (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 88825
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: COVID-19
Keywords: Booster dose Moderna and Pfizer; mRNA vaccine; monovalent, bivalent
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine; 2019-nCoV Vaccine mRNA-1273; BNT162b5

STUDY DESIGN:
Intervention Model Description: Study participants who have received two doses of either Pfizer or Astrazena vaccine as their primary vaccine and a standard dose of Pfizer for their booster will be randomised into one of four groups. The four groups consist of a standard dose of either the monovalent or bivalent Pfizer or Moderna vaccine.
Who Masked: Participant, Investigator
Masking Description: The participants and those evaluating reactogenicity will be blinded to the vaccine allocation for the first 7 days following vaccination. After that, both clinical investigators and participants will be aware of their investigational product. Laboratory staff will remain blinded to the investigational product.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Monovalent Pfizer-BioNTech(BNT162b2): Pfizer-BioNTech(BNT162b2)-Pfizer-BioNTech(BNT162b2) (Active Comparator): Participants who received Pfizer-BioNTech(BNT162b2) as primary series and Pfizer-BioNTech(BNT162b2) as first booster will receive a second booster dose of:
  Biological/Vaccine: Tozinameran - Monovalent Tozinamrean is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cell-free in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Interventions: Biological: Tozinameran
- Monovalent Moderna(mRNA-1273, Spikevax®): Pfizer-BioNTech(BNT162b2)-Pfizer-BioNTech(BNT162b2) (Active Comparator): Participants who received Pfizer-BioNTech(BNT162b2) as primary series and Pfizer-BioNTech(BNT162b2) as first booster will receive a second booster dose of:
  Biological/Vaccine: Elasomeran - Monovalent Elasomeran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cell-free in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of SARS-CoV-2).
  Interventions: Biological: Elasomeran
- Monovalent Pfizer-BioNTech(BNT162b2): AstraZeneca(ChAdOx1, Vaxzevria®)-Pfizer-BioNTech(BNT162b2) (Active Comparator): Participants who received AstraZeneca (ChAdOx1, or Vaxzevria®) as primary series and Pfizer-BioNTech (BNT162b2) as first booster will received a second booster dose of:
  Biological/Vaccine: Tozinameran - Monovalent Tozinamrean is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cell-free in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Interventions: Biological: Tozinameran
- Monovalent Moderna(mRNA-1273, Spikevax®):AstraZeneca(ChAdOx1, Vaxzevria®)-Pfizer-BioNTech(BNT162b2) (Active Comparator): Participants who received AstraZeneca (ChAdOx1, or Vaxzevria®) as primary series and Pfizer-BioNTech (BNT162b2) as first booster will received a second booster dose of:
  Biological/Vaccine: Elasomeran - Monovalent Elasomeran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cell-free in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of SARS-CoV-2).
  Interventions: Biological: Elasomeran
- Bivalent Pfizer-BioNTech (BNT162b2 OMI): Pfizer-BioNTech(BNT162b2)-Pfizer-BioNTech(BNT162b2) (Active Comparator): Participants who received Pfizer-BioNTech(BNT162b2) as primary series and Pfizer-BioNTech(BNT162b2) as first booster will receive a second booster dose of:
  Biological/Vaccine: Pfizer-BioNTech, BNT162b2 OMI - bivalent Pfizer-BioNTech bivalent COVID-19 vaccine contains ancestral BNT162b2 and Omicron variant BNT162b2 Omi (BA.1). The Pfizer-BioNTech COVID-19 vaccine, BNT162b2, encodes a P2 mutant spike protein and is formulated as an RNA-lipid nanoparticle (LNP) of nucleoside-modified mRNA (modRNA).
  Interventions: Biological: Bivalent Pfizer-BioNTech
- Bivalent Moderna (mRNA-1273.214): Pfizer-BioNTech(BNT162b2)-Pfizer-BioNTech(BNT162b2) (Active Comparator): Participants who received Pfizer-BioNTech(BNT162b2) as primary series and Pfizer-BioNTech(BNT162b2) as first booster will receive a second booster dose of:
  Biological/Vaccine: Moderna, mRNA-1273.214 - bivalent The Moderna bivalent vaccine (mRNA-1273.214) encodes the prefusion stabilized S protein of SARS-CoV-2 formulated in RNA-lipid nanoparticles composed of 4 lipids and 1-monomethoxypolyethyleneglycol-2, 3-dimyristylglycerol with polyethylene glycol. 25μg of each mRNA sequence that encode the prefusion stabilized spike glycoproteins of the ancestral SARS-CoV-2 (Wuhan-Hu-1) and the Omicron variant (B.1.1.529 [BA.1]).
  Interventions: Biological: Bivalent Moderna
- Bivalent Pfizer-BioNTech (BNT162b2): AstraZeneca(ChAdOx1, Vaxzevria®)-Pfizer-BioNTech(BNT162b2) (Active Comparator): Participants who received AstraZeneca (ChAdOx1-S, or Vaxzevria®) as primary series and Pfizer-BioNTech (BNT162b2) as first booster will received a second booster dose of:
  Biological/Vaccine: Pfizer-BioNTech, BNT162b2 OMI - bivalent Pfizer-BioNTech bivalent COVID-19 vaccine contains ancestral BNT162b2 and Omicron variant BNT162b2 Omi (BA.1). The Pfizer-BioNTech COVID-19 vaccine, BNT162b2, encodes a P2 mutant spike protein and is formulated as an RNA-lipid nanoparticle of nucleoside-modified mRNA.
  Interventions: Biological: Bivalent Pfizer-BioNTech
- Bivalent Moderna (mRNA-1273.214): AstraZeneca(ChAdOx1, Vaxzevria®)-Pfizer-BioNTech(BNT162b2) (Active Comparator): Participants who received AstraZeneca (ChAdOx1-S, or Vaxzevria®) as primary series and Pfizer-BioNTech (BNT162b2) as first booster will received a second booster dose of:
  Biological/Vaccine: Moderna, mRNA-1273.214 - bivalent The Moderna bivalent vaccine (mRNA-1273.214) encodes the prefusion stabilized S protein of SARS-CoV-2 formulated in RNA-lipid nanoparticles composed of 4 lipids and 1-monomethoxypolyethyleneglycol-2, 3-dimyristylglycerol with polyethylene glycol. 25μg of each mRNA sequence that encode the prefusion stabilized spike glycoproteins of the ancestral SARS-CoV-2 (Wuhan-Hu-1) and the Omicron variant (B.1.1.529 [BA.1]).
  Interventions: Biological: Bivalent Moderna

INTERVENTIONS:
Biological: Tozinameran — A single standard dose (30mcg) will be administered on day 0 of the study.
  Other Names: BNT162b2, Pfizer-BioNTech, Comirnaty
  Arms: Monovalent Pfizer-BioNTech(BNT162b2): Pfizer-BioNTech(BNT162b2)-Pfizer-BioNTech(BNT162b2)
Biological: Elasomeran — A single standard dose (50mcg) of the intervention will be administered on day 0 of the study.
  Other Names: mRNA-1273, Spikevax, Moderna
  Arms: Monovalent Moderna(mRNA-1273, Spikevax®): Pfizer-BioNTech(BNT162b2)-Pfizer-BioNTech(BNT162b2)
Biological: Tozinameran — A single standard dose (30mcg) will be administered on day 0 of the study.
  Other Names: BNT162b2, Pfizer-BioNTech, Comirnaty
  Arms: Monovalent Pfizer-BioNTech(BNT162b2): AstraZeneca(ChAdOx1, Vaxzevria®)-Pfizer-BioNTech(BNT162b2)
Biological: Elasomeran — A single standard dose (50mcg) of the intervention will be administered on day 0 of the study.
  Other Names: mRNA-1273, Spikevax, Moderna
  Arms: Monovalent Moderna(mRNA-1273, Spikevax®):AstraZeneca(ChAdOx1, Vaxzevria®)-Pfizer-BioNTech(BNT162b2)
Biological: Bivalent Pfizer-BioNTech — A single standard dose (BNT162b2 15μg +BNT162b2 OMI 15μg) will be administered on day 0 of the study.
  Other Names: BNT162b2 + BNT162b2 OMI
  Arms: Bivalent Pfizer-BioNTech (BNT162b2 OMI): Pfizer-BioNTech(BNT162b2)-Pfizer-BioNTech(BNT162b2)
Biological: Bivalent Moderna — A single standard dose (BNT162b2 15μg + BNT162b2 OMI 15μg)will be administered on day 0 of the study.
  Other Names: mRNA-1273.214 +B.1.1.529 OMI
  Arms: Bivalent Moderna (mRNA-1273.214): Pfizer-BioNTech(BNT162b2)-Pfizer-BioNTech(BNT162b2)
Biological: Bivalent Pfizer-BioNTech — A single standard dose (BNT162b2 15μg + BNT162b2 OMI 15μg) will be administered on day 0 of the study.
  Other Names: BNT162b2 + BNT162b2 OMI
  Arms: Bivalent Pfizer-BioNTech (BNT162b2): AstraZeneca(ChAdOx1, Vaxzevria®)-Pfizer-BioNTech(BNT162b2)
Biological: Bivalent Moderna — A single standard dose (BNT162b2 15μg +BNT162b2 OMI 15μg) will be administered on day 0 of the study.
  Other Names: mRNA-1273.214 +B.1.1.529 OMI
  Arms: Bivalent Moderna (mRNA-1273.214): AstraZeneca(ChAdOx1, Vaxzevria®)-Pfizer-BioNTech(BNT162b2)

SUMMARY:
This clinical trial will be a blinded, randomised study to determine the safety, reactogenicity, and immunogenicity of a second booster dose of SARS-CoV-2 vaccines in adults enrolled over two consecutive stages. Stage 1 will commence at the time of study approval and transition to stage 2 once bivalent vaccines are approved and available in Australia.

DETAILED DESCRIPTION:
Participants will be adults aged 18 years or older who have been previously primed with two doses of either Pfizer-BioNTech (BNT162b2, or Comirnaty®) or AstraZeneca (ChAdOx1-S, or Vaxzevria®) and boosted at least 3 months earlier with Pfizer BioNTech vaccine (30µg). There will be no upper age limit. Participants will be recruited from the Murdoch Children's Research Institute, the Royal Children's Hospital (RCH), the Peter Doherty Research Institute, and, if necessary, the greater Melbourne area. Ideally, 100 participants will be recruited per group unless bivalent Omicron-specific vaccines are introduced before this target is reached for monovalent ancestral vaccines. There will be 800 participants in total. Procedures will be implemented to ensure participants of all ages (aged 18 and above) are included and that there is an even age distribution in each group (<50 and ≥50 years).

ELIGIBILITY:
Inclusion Criteria:

1. Have completed a primary schedule of two doses of Pfizer-BioNTech or AstraZeneca vaccines and received a booster of Pfizer-BioNTech vaccine (30µg) at least 3 months earlier.
2. No confirmed SARS-CoV-2 infection on PCR or RAT within the last 3 months.
3. Willing and able to give written informed consent.
4. Aged 18 years or above.
5. Willing to complete the follow-up requirements of the study.

Exclusion Criteria:

1. Currently receiving immunosuppressive medication or anti-cancer chemotherapy.
2. Known HIV infection.
3. Congenital immune deficiency syndrome.
4. Received immunoglobulin or other blood products in the three months prior to potential study booster vaccination.
5. Study staff and their relatives.
6. Have a history of a severe allergic reaction to any COVID-19 vaccines or have a medical exemption to receiving further COVID-19 vaccines.
7. Cannot read or understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 specific Immunoglobulin (Ig)G antibodies at 28-days post booster vaccination | 28-days post booster vaccination
  Serum samples collected at 28-days post booster vaccination from all groups will be evaluated for SARS-CoV-2 specific IgG antibodies using the commercial Euroimmun S1 IgG ELISA. Data will be reported as binding antibody units/mL and presented as geometric mean concentration and 95% confidence intervals
Total incidence of solicited reactions (systemic and local) | Total incidence of solicited reactions will be measured for 7 days post booster vaccination
  Questionnaire to document solicited reactions is developed specifically for this study. Data will be reported as the proportion of participants who report by each intervention arm. Solicited reactions such as pain, tenderness, erythema/redness, induration/swelling, fever, nausea/vomiting, headache, fatigue/malaise, myalgia, arthralgia will be collected from the participants 7 days post-vaccination.

SECONDARY OUTCOMES:
SARS-CoV-2 specific IgG antibodies at baseline (pre booster), and 6-months post booster vaccination | Baseline (pre booster), and 6-months post booster vaccination
  Serum samples collected at baseline (pre booster), and 6-months post booster vaccination from all groups will be evaluated for SARS-CoV-2 specific IgG antibodies using the commercial Euroimmun S1 IgG ELISA . Data will be reported as binding antibody units/mL and presented as geometric mean concentration and 95% confidence intervals
SARS-CoV-2 specific neutralising antibodies at baseline (pre booster), 28 days and 6-months post booster vaccination measured by surrogate virus neutralization test (sVNT) | Baseline (pre booster), 28 days and 6 months post booster vaccination
  Serum samples collected at baseline (pre booster), 28 days- and 6-months post booster vaccination from all groups will be evaluated for SARS-CoV-2 specific neutralising antibodies using the GenScript® cPass surrogate virus neutralization test (sVNT) for both wild-type and Omicron variant. Neutralising antibody response will be reported as percentage (%) inhibition of receptor binding domain-angiotensin-converting enzyme 2 (RBD-ACE2) binding relative to a positive control.
SARS-CoV-2 specific neutralising antibodies at baseline (pre booster), 28 days and 6- months post booster vaccination measured by SARS-CoV-2 microneutralisation assay | Baseline (pre booster), 28 days-, and 6-months post booster vaccination
  A subset of samples from all timepoints will be assessed using a SARS-CoV-2 microneutralisation assay to both the wild type (vaccine) strain and for two SARS-CoV-2 Variants of concern. Neutralizing antibody will be reported as endpoint titre.
Interferon gamma (IFNγ) concentrations in International Units (IU)/mL | Baseline (pre booster), 28 days-, and 6-months post booster vaccination
  Interferon gamma (IFNγ) concentrations as a measurement of cellular immunity will be assessed on a subset (40%) of the participants from each group. QuantiFERON Human IFN-γ SARS-CoV-2 (Qiagen) will be used to stimulate IFN-γ production in peripheral blood mononuclear cells (PBMCs) and then IFN-γ production will be measured using ELISA. Data will be presented as geometric mean concentration (GMC) and 95% confidence intervals (CI).
Number of IFNγ producing cells/million PBMCs | Baseline (pre booster), 28 days-, and 6-months post booster vaccination
  IFNγ producing cells as a measurement of cellular immunity will be assessed on a subset (40%) of the participants from each group. IFN-γ Enzyme-Linked ImmunoSpot (Elispot) assay will be performed on isolated peripheral blood mononuclear cells (PBMCs). Data will be reported as number of IFNγ producing cells/million and presented using means and 95% confidence intervals.
Frequency of cytokine-expressing T cells | Baseline (pre booster), 28 days-, and 6-months post booster vaccination
  Frequency of cytokine-expressing T cells will be assessed on a subset (40%) of participants using Flow cytometry (intracellular staining) on PBMCs samples. Data will be reported as frequency (%) of cytokine-expressing T cells presented as means and 95% CI.
Cytokine concentrations following PBMCs stimulation | Baseline (pre booster), 28 days and 6-months post booster vaccination
  Cytokine concentrations following PBMCs stimulation will be assessed on a subset (40%) of participants using multiplex cytokine assays.Data will be reported as cytokine concentrations in pg/ml and presented as GMC and 95% CI.
Incidence of unsolicited adverse events (AE) | 28 days-post booster vaccination
  All unsolicited AE will be collected for 28 days post booster vaccination. Data will be presented as proportion of participants who report unsolicited AE.
Incidence of medically attended adverse events (AE) | 3 months post booster vaccination
  Participants with medically attended AE will be collected for 3 months post booster vaccination. Data will be presented as proportion of participants who report unsolicited AE.
Incidence of serious adverse events (SAE) | 6 months post booster vaccination
  SAE will be collected throughout the follow-up period of 6 months post booster vaccination. Data will be presented as a proportion of participants who report unsolicited SAE.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Mulholland, MD/Prof, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Royal Children's Hospital, Murdoch Children's Research Institute, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified data to ethically approved studies in cases where participants have indicated on the consent form that they consent to the use of their data and where consistent with terms of collaboration agreements.
Supporting Information: Study Protocol, ICF
Time Frame: Individual participant data (IPD) sharing plans in development
Access Criteria: In development

REFERENCES:
- [Derived] Mazarakis N, Toh ZQ, Neal E, Bright K, Luu S, Quah L, Ng YY, Nguyen C, Hart J, Do LAH, Rudel A, Dassanayake S, Higgins RA, Ong DS, Justice F, Moore KA, Watts E, Mahanty S, Subbarao K, Mulholland K, von Mollendorf C, Licciardi PV. The immunogenicity, reactogenicity, and safety of a bivalent mRNA or protein COVID-19 vaccine given as a fourth dose. J Infect. 2025 Mar;90(3):106447. doi: 10.1016/j.jinf.2025.106447. Epub 2025 Feb 18. PMID 39978439
- See also: World Health Organization. Interim statement on the use of additional booster doses of Emergency Use Listed mRNA vaccines against COVID-19 2022 — https://www.who.int/news/item/17-05-2022-interim-statement-on-the-use-of-additional-booster-doses-of-emergency-use-listed-mrna-vaccines-against-covid-19
- See also: US Food and Drug Administration (FDA). Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials 2007 — https://www.fda.gov/media/73679/download
- See also: International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use. Addendum on Estimands and Sensitivity Analysis in Clinical Trials to the Guideline on Statistical Principles for Clinical Trials 2019 — https://database.ich.org/sites/default/files/E9-R1_Step4_Guideline_2019_1203.pdf